CLINICAL TRIAL: NCT01812122
Title: Effects of Vildagliptine and Glimepiride on Glycemic Variability and Cardiovascular Parameters in Patients With Type 2 Diabetes by CGMS
Brief Title: Effects of Vildagliptine and Glimepiride on Glucose Variability
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hye Seung Jung, Assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CGMS_SU_Gliptin
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride; Vildagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glimepiride (Experimental): Starting with Glimepiride. After 3 month, switching to vildagliptin.
  Interventions: Drug: Glimepiride; Drug: Vildagliptin
- Vildagliptin (Experimental): Starting with vildagliptin. After 3 month, switching to Glimepiride.
  Interventions: Drug: Glimepiride; Drug: Vildagliptin

INTERVENTIONS:
Drug: Glimepiride
Drug: Vildagliptin

SUMMARY:
The purpose of this study is to analyze the differences of blood sugar level and glycemic variability between sulfonylurea and DPP-4 inhibitor groups applying CGMS for a chosen number of type 2 DM patients. The investigators also reveal influences of each drugs on cardiovascular risk factors by measuring related biomarkers.

DETAILED DESCRIPTION:
We enroll patients with type 2 DM with uncontrolled glucose level on Metformin monotherapy over 1000mg /day (HbA1C over 7%).

Before drug administration, we conduct basal lab study including CGMS. After 3 month of random administration of vildagliptin or glimepiride, we check CGMS, glucose levels, CV biomarkers, and estimate hypoglycemic index. We replace with the other drug for 3 months, and then conduct the same measurements. No wash-out period is necessary since result variables are measured after the 3 months of administration for a different drug.

ELIGIBILITY:
Inclusion Criteria:

* with type 2 DM
* with uncontrolled glucose level on Metformin monotherapy over 1000mg /day (HbA1C over 7%). Provided that the tolerance for metformin is poor, enrollment of patients with lower dose of metfomrin is open.
* who have never been prescribed with test drugs, sulfonylurea or DPP-4 inhibitor/GLP-1 analogue in 3 months
* who can be applied with CGMS

Exclusion Criteria:

* who has liver function abnormality or renal function abnormality
* who has any kind of diseases, operations, medical treatments that can affect glucose levels

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-03; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Glycemic variability index | before and after 3 months of each drug administration
Cardiovascular disease risk factor | before and after 3 months of each drug administration

SECONDARY OUTCOMES:
glucose profile and lipid profile | before and after 3 months of each drug administration
hypoglycemic index | before and after 3 months of each drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Hye Seung Jung, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea